CLINICAL TRIAL: NCT06687746
Title: Multi-Country Evaluation of Bili-ruler, a Low-cost Icterometer for Screening of Jaundice in Newborns
Brief Title: Evaluation of Bili-ruler, a Low-cost, Plastic Icterometer for Community-based Screening of Jaundice in Newborns
Status: Active, not recruiting | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: Kenya Medical Research Institute (Other); University of North Carolina, Chapel Hill (Other); Kintampo Health Research Centre, Ghana (Other); Aga Khan University (Other); Christian Medical College, Vellore, India (Other); Society for Applied Studies (Other); Liverpool School of Tropical Medicine, United Kingdom (Unknown); University of Ghana (Other); University of North Carolina Global Project Zambia (Unknown)
Responsible Party: Principal Investigator, Emily Smith, Principal Investigator, George Washington University
Other Study IDs: BILIRULER2024
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Jaundice, Neonatal; Neonatal Diseases and Abnormalities; Neonatal Hyperbilirubinemia; Screening Tool; Screening
Keywords: Hyperbilirubinemia; Jaundice; Neonatology; Universal Screening; Cohort Study; Icterometry
MeSH Terms: conditions — Jaundice, Neonatal; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Hyperbilirubinemia, Neonatal; Hyperbilirubinemia; Jaundice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Pakistan Cohort: Infants born to PRISMA-enrolled mothers in the Pakistan catchment area
  Interventions: Device: Bili-ruler
- Kenya Cohort: Infants born to PRISMA-enrolled mothers in the Kenya catchment area
  Interventions: Device: Bili-ruler
- Ghana Cohort: Infants born to PRISMA-enrolled mothers in the Ghana catchment area
  Interventions: Device: Bili-ruler
- Zambia Cohort: Infants born to PRISMA-enrolled mothers in the Zambia catchment area
  Interventions: Device: Bili-ruler
- Vellore, India Cohort: Infants born to PRISMA-enrolled mothers in the Vellore, India catchment area
  Interventions: Device: Bili-ruler
- Hodal, India Cohort: Infants born to PRISMA-enrolled mothers in the Hodal, India catchment area
  Interventions: Device: Bili-ruler

INTERVENTIONS:
Device: Bili-ruler — The noninvasive test will be conducted by aligning the bili-ruler with the infant's nose and choosing the color on the ruler which most closely matches the yellow discoloration on the skin.

SUMMARY:
Newborn jaundice, or accumulation of bilirubin molecules in blood, affects 60-80% of newborns and, in severe cases, places newborns at risk of brain damage and death. Universal screening of all newborn for jaundice ensures that at-risk newborns are identified and treated early. The bili-ruler is a low-cost ($10) plastic icterometer which could enable accurate and timely identification of jaundice in diverse settings.

The objective of this study is to evaluate the ability of bili-ruler to identify jaundiced newborns in their first week of life, compared to traditional methods of jaundice screening: visual inspection and transcutaneous bilirubinometry.

DETAILED DESCRIPTION:
Neonatal jaundice, or accumulation of bilirubin molecules in blood, places newborns at risk of brain damage and death. Hyperbilirubinemia, or severe bilirubin levels above approximately 15 mg/dL, is a secondary outcome in the PRISMA MNH study. Newborn jaundice accounted for 13.09 deaths per 100,000 in 2016, and the burden is highest in South Asia and sub-Saharan Africa, where neonatal jaundice is the 7th and 8th leading cause of newborn mortality, respectively. Universal screening is recommended, but the standard of care, visual inspection of the skin and sclera, has a low sensitivity of 42%. Transcutaneous bilirubinometers are promising noninvasive, handheld tools, but they are expensive (> $3000) and inaccurate in newborns with darker skin. In low-and-middle-income countries, as well as in rural settings, guardians and clinicians often fail to identify at-risk newborns due to a lack of appropriate, affordable, and accurate screening tools. The bili-ruler is a $10 ruler with six shades of yellow, which could enable jaundice screening with high sensitivity in diverse settings such as homes, mobile clinics, and rural areas.

In this study, we will evaluate jaundice in newborns using three noninvasive techniques: bili-ruler, visual inspection, and transcutaneous bilirubinometry (a handheld device). The goals are to determine whether the six bili-ruler shades of yellow can be accurately correlated with bilirubin levels measured by a transcutaneous device, as well as to evaluate whether many users from various backgrounds can easily use bili-ruler to obtain comparable measurements. Additionally, limited evidence exists on the progression of jaundice and the performance of noninvasive screening tools in premature newborns and in newborns with various skin tones, especially darker skin tones. We seek to address this gap by utilizing an existing multi-site, international collaboration (the Pregnancy Risk, Infant Surveillance, and Measurement Alliance, or PRISMA) and enrolling large, diverse study populations. This study is nested in the PRISMA Maternal and Newborn Health (MNH) study, which is an open-cohort study that assesses pregnancy risk factors and associated maternal and infant outcomes in six study sites in five countries. All six study sites, located in Ghana, Zambia, Kenya, Pakistan, and India, will participate and collect bilirubin and jaundice-related data at four time points (0-3, 3-5, 5-7, and 7-14 days of life). The investigators will evaluate agreement between the three methods and agreement between bili-ruler measurements taken by two independent users. The investigators will additionally evaluate the impact of gestational age and skin tone on the accuracy of bili-ruler. Finally, the investigators will assess factors that influence bilirubin measurements.

ELIGIBILITY:
Inclusion Criteria:

* All infants who are born to PRISMA enrolled mothers will be eligible for this study.

Exclusion Criteria:

* Presence of skin lesions, abnormalities, etc on the baby's nose, face, and ears, which could interfere with bilirubin measurement, as determined by research staff.

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants who are born to mothers in the catchment areas covered by PRISMA study sites
Sampling Method: Non-Probability Sample
Enrollment: 5400 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Bilirubin | 0-3 days of life
  Bilirubin levels will be assessed using Bili-ruler and a transcutaneous bilirubinometer (the Mennin Medical BiliCare device) at 0-3 days of life.
Bilirubin | 3-5 days of life
  Bilirubin levels will be assessed using Bili-ruler and a transcutaneous bilirubinometer (the Mennin Medical BiliCare device) at 3-5 days of life.
Bilirubin | 5-7 days of life
  Bilirubin levels will be assessed using Bili-ruler and a transcutaneous bilirubinometer (the Mennin Medical BiliCare device) at 5-7 days of life.

SECONDARY OUTCOMES:
Jaundice | 0-3 days of life
  Jaundice will be evaluated using visual inspection of the skin and sclera of the newborn. We will define 'jaundice' as the presence of yellow discoloration on the newborn's forehead, and we will define 'severe jaundice' as the presence of yellow discoloration on the palms/soles.
Jaundice | 3-5 days of life
  Jaundice will be evaluated using visual inspection of the skin and sclera of the newborn. We will define 'jaundice' as the presence of yellow discoloration on the newborn's forehead, and we will define 'severe jaundice' as the presence of yellow discoloration on the palms/soles.
Jaundice | 5-7 days of life
  Jaundice will be evaluated using visual inspection of the skin and sclera of the newborn. We will define 'jaundice' as the presence of yellow discoloration on the newborn's forehead, and we will define 'severe jaundice' as the presence of yellow discoloration on the palms/soles.

CONTACTS AND LOCATIONS:
Locations (6):
- Kintampo Health Research Centre, Kintampo, Ghana, Ghana
- India (2):
  - Society for Applied Studies (SAS), Hodal, India
  - Christian Medical College (CMC), Vellore, India
- Kenya Medical Research Institute - Center for Global Health Research, Kisumu, Kenya, Kenya
- Aga Khan University, Karachi, Pakistan, Pakistan
- University of North Carolina - Global Projects Zambia, Lusaka, Zambia, Zambia

IPD SHARING:
Plan to Share IPD: No